CLINICAL TRIAL: NCT00096486
Title: A Phase I/II Trial of Fixed Doses of Daily Gefitinib With Escalating Doses of Daily RAD001 in Advanced Non-Small Cell Lung Cancer
Brief Title: Gefitinib and Everolimus in Treating Patients With Stage IIIB or Stage IV or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-033; MSKCC-04033
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Everolimus; Gefitinib

ARMS (1):
- Gefitinib and Everolimus (RAD001) (Experimental): Phase I: Patients receive oral everolimus once on day 1. Beginning on day 8, patients receive oral gefitinib once daily. Beginning on day 22, patients receive oral everolimus once daily. Both drugs are then given concurrently for the rest of the treatment. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of everolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.
  * Phase II: Patients receive oral everolimus at the MTD determined in phase I and oral gefitinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus; Drug: gefitinib

INTERVENTIONS:
Drug: everolimus
Drug: gefitinib

SUMMARY:
RATIONALE: Gefitinib and everolimus may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving gefitinib together with everolimus may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects, best way to give, and best dose of giving gefitinib with everolimus and to see how well it works in treating patients with stage IIIB or stage IV or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of everolimus when administered with gefitinib in patients with stage IIIB or IV or recurrent non-small cell lung cancer. (Phase I)
* Determine the efficacy of this regimen in these patients. (Phase II)

Secondary

* Assess the pharmacokinetics of everolimus, alone and in combination with gefitinib, in these patients. (Phase I)

OUTLINE: This is an open-label, phase I, dose-escalation study of everolimus followed by a phase II study.

* Phase I: Patients receive oral everolimus once on day 1. Beginning on day 8, patients receive oral gefitinib once daily. Beginning on day 22, patients receive oral everolimus once daily. Both drugs are then given concurrently for the rest of the treatment. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of everolimus until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experiences dose-limiting toxicity.

* Phase II: Patients receive oral everolimus at the MTD determined in phase I and oral gefitinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC) meeting 1 of the following stage criteria:

  * Stage IIIB (unresectable, with malignant pleural or pericardial effusion)
  * Stage IV disease
  * Recurrent disease
* Measurable or evaluable indicator lesions
* Progressive disease after receiving ≥ 1 prior chemotherapy regimen that included cisplatin or carboplatin and docetaxel
* No uncontrolled brain or leptomeningeal metastases

  * Must not require concurrent glucocorticoids for control of metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100% OR
* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No congestive heart failure
* No New York Heart Association class III or IV heart disease
* No unstable angina

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No severe infection
* No severe malnutrition
* No other serious medical illness
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer or carcinoma of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy
* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* No prior conventional chemotherapy for metastatic or recurrent NSCLC (phase II only)
* At least 4 weeks since prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent oral steroids for management of skin toxicity

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* At least 4 weeks since prior major surgery
* No concurrent surgery for an identifiable lesion

Other

* Recovered from all prior therapy
* No prior gefitinib, erlotinib, or other epidermal growth factor tyrosine kinase inhibitor
* No concurrent cytotoxic therapy (e.g., methotrexate for rheumatoid arthritis)
* No other concurrent oncolytic agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2004-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent A. Miller, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Price KA, Azzoli CG, Krug LM, Pietanza MC, Rizvi NA, Pao W, Kris MG, Riely GJ, Heelan RT, Arcila ME, Miller VA. Phase II trial of gefitinib and everolimus in advanced non-small cell lung cancer. J Thorac Oncol. 2010 Oct;5(10):1623-9. doi: 10.1097/JTO.0b013e3181ec1531. PMID 20871262

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: RAD001 10 mg, Gefitinib 250 mg: Phase I: RAD001 10 mg, Gefitinib 250 mg
- Phase I: RAD001 5 mg, Gefitinib 250 mg: Phase I: RAD001 5 mg, Gefitinib 250 mg
- Phase II: Cohort I no Prior Conventional Chemotherapy: Phase II: Cohort I no prior conventional chemotherapy
- Phase II: Cohort II One or More Prior Chemotherapy: Phase II: Cohort II one or more prior chemotherapy
Period: Overall Study
Arm/Group | Phase I: RAD001 10 mg, Gefitinib 250 mg | Phase I: RAD001 5 mg, Gefitinib 250 mg | Phase II: Cohort I no Prior Conventional Chemotherapy | Phase II: Cohort II One or More Prior Chemotherapy
Started | 4 | 6 | 26 | 38
Completed | 4 | 6 | 24 | 36
Not Completed | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1
Not completed — Not Treated | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: RAD001 10 mg, Gefitinib 250 mg | Phase I: RAD001 5 mg, Gefitinib 250 mg | Phase II: Cohort I no Prior Conventional Chemotherapy | Phase II: Cohort II One or More Prior Chemotherapy | Total
Number analyzed (Participants) | 4 | 6 | 26 | 38 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 8 | 23 | 36
  >=65 years | 3 | 2 | 18 | 15 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 10 | 22 | 36
  Male | 2 | 4 | 16 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Determine efficacy of the combination oral daily gefitinib and oral daily RAD001 in patients with advanced NSCLC. Response and progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Phase I: RAD001 10 mg, Gefitinib 250 mg | Phase I: RAD001 5 mg, Gefitinib 250 mg | Phase II: Cohort I no Prior Conventional Chemotherapy | Phase II: Cohort II One or More Prior Chemotherapy
Number analyzed (Participants) | 4 | 6 | 24 | 36
participants
  Partial Response (PR) | 1 | 1 | 3 | 2
  Stable Disease (SD) | 1 | 1 | 9 | 15
  Progression of Disease (POD) | 1 | 4 | 11 | 18
  Not Evaluable/ Evaluable for Toxicity Only | 1 | 0 | 1 | 1

ADVERSE EVENTS:
Arm/Group | Phase I: RAD001 10 mg, Gefitinib 250 mg | Phase I: RAD001 5 mg, Gefitinib 250 mg | Phase II: Cohort I no Prior Conventional Chemotherapy | Phase II: Cohort II One or More Prior Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/6 | 5/26 | 15/38
Other Adverse Events (participants affected / at risk) | 3/4 | 5/6 | 20/26 | 28/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: RAD001 10 mg, Gefitinib 250 mg (N=4) | Phase I: RAD001 5 mg, Gefitinib 250 mg (N=6) | Phase II: Cohort I no Prior Conventional Chemotherapy (N=26) | Phase II: Cohort II One or More Prior Chemotherapy (N=38)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death not associated with CTCAE term- Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death not associated with CTCAE term- Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death not associated with CTCAE term-Disease prog NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness - Whole body/general (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain - Abdomen (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Back (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain - Chest wall (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Extremity-limb (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Secondary malignancy-possibly related to cancer treatment specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (fainting) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: RAD001 10 mg, Gefitinib 250 mg (N=4) | Phase I: RAD001 5 mg, Gefitinib 250 mg (N=6) | Phase II: Cohort I no Prior Conventional Chemotherapy (N=26) | Phase II: Cohort II One or More Prior Chemotherapy (N=38)
Anorexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (6) | 4 (8)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 3 (3) | 7 (7) | 15 (15)
INR (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Mucositis (Clincal exam)- Oral cavity (General disorders) | 1 (2) | 0 (0) | 13 (24) | 14 (16)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 8 (8) | 14 (15)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Mucositis (symptoms)- Oral cavity (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes